CLINICAL TRIAL: NCT00700713
Title: Antibody Persistence and Booster Dose Response in Subjects Who Received Menactra® (Meningococcal [Groups A, C, Y, and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) Three Years Earlier in Study MTA26
Brief Title: Antibody Persistence and Booster Dose Response in Subjects Who Received Menactra® Three Years Earlier in Study MTA26
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA62
Record Dates: First submitted 2008-05-07; First posted 2008-06-19 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Meningitis; Meningococcemia
Keywords: Meningitis; Meningococcemia; Neisseria meningitidis; Menactra®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- One-Dose Menactra Group (Experimental): Participants received one dose of Menactra® in Study MTA26
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate
- Two-Dose Menactra Group (Experimental): Participants received two doses of Menactra® in Study MTA26
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate
- Menactra vaccine-naïve Group (Active Comparator): Participants had never received Menactra® vaccine.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate

INTERVENTIONS:
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate — 0.5 mL, IM
  Other Names: Menactra®
  Arms: One-Dose Menactra Group
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate — 0.5 mL, IM
  Other Names: Menactra®
  Arms: Two-Dose Menactra Group
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate — 0.5 mL, IM
  Other Names: Menactra®
  Arms: Menactra vaccine-naïve Group

SUMMARY:
Study will evaluate the persistence of antibodies approximately three years after an initial dose of Menactra® vaccine in toddlers who participated in study MTA26 (NCT00643916) and age-matched Menactra naive participants.

Objectives:

* To assess the persistence of antibody responses three years after one or two doses of Menactra® vaccine in subjects who participated in study MTA26.
* To describe the antibody responses to a single dose of Menactra® vaccine in subjects who had previously received one or two doses of Menactra® vaccine and in Menactra® vaccine-naïve subjects.
* To describe the safety profile of a single dose of Menactra® vaccine in subjects.

DETAILED DESCRIPTION:
Subjects that received Menactra® vaccine in study MTA26 (NCT00643916) and age-matched Menactra naive participants will receive a single dose of Menactra® on Day 0. They will be evaluated for immunogenicity and safety post-vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Subjects received one or two doses of Menactra® vaccine in study MTA26 and provided a blood sample after the last dose received
* At 3 to < 6 years of age and were never vaccinated against meningococcal disease (with either the study vaccine or another vaccine).
* Informed consent form signed and dated by the parent(s) or another legally acceptable representative.
* Subject and parent/legal guardian able to attend all scheduled visits and comply with all study procedures.

Exclusion Criteria :

* Participation in the active (i.e., treatment) portion of another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first study vaccination
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known or suspected systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the study vaccine or to a product containing any of the substances present in the study vaccine.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator.
* Received blood or blood-derived products in the past 3 months.
* Received any vaccine (other than desensitization therapy for allergies or influenza vaccine within 2 weeks before vaccination) in the 4 weeks preceding the first study vaccination.
* Planned receipt of any vaccine within the 4 weeks following the study vaccination.
* Known human immunodeficiency virus (HIV), hepatitis B surface antigen (HBs antigen), or hepatitis C seropositivity.
* History of invasive meningococcal infection (confirmed either clinically, serologically, or microbiologically).
* Thrombocytopenia, coagulation disorder, or anticoagulant use in the 3 weeks preceding inclusion contraindicating intramuscular (IM) vaccination.
* Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to any of the trial blood draws.
* Personal or family history of Guillain-Barré Syndrome (GBS).
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (12):
- United States (12):
  - Marietta, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Annapolis, Maryland
  - Frederick, Maryland
  - Woburn, Massachusetts
  - Greenville, Pennsylvania
  - Harleysville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Kingsport, Tennessee
  - Layton, Utah
  - Provo, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 17 June 2008 to 01 October 2008 at 13 clinical centers in the United States.
Pre-assignment Details: A total of 181 participants who met all inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Menactra-naïve Group: Participants had never received Menactra® vaccine.
Period: Overall Study
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group
Started | 48 | 66 | 67
Completed | 47 | 66 | 65
Not Completed | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group | Total
Number analyzed (Participants) | 48 | 66 | 67 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 66 | 67 | 181
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 57.4 (2.89) | 51.6 (1.96) | 52.5 (11.8) | 53.4 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 38 | 22 | 80
  Male | 28 | 28 | 45 | 101
Region of Enrollment [Number; unit: Participants]
  United States | 48 | 66 | 67 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Meningococcal Serogroups A, C, Y, and W-135 Bactericidal Antibody Titers ≥ 1:4 and ≥ 1:8 Before and Following Vaccination With Menactra®
Description: Antibody titers to meningococcal serogroups A, C, Y, and W-135 were measured by serum bactericidal assay using human complement (SBA-HC). Bactericidal antibody persistence to meningococcal serogroups was defined as as pre-vaccination titers of ≥1:4 and ≥1:8. Booster response to a single Menactra vaccine dose was defined as antibody titers of ≥1:4 and ≥1:8 30 days post-booster vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Meningococcal serogroups A, C, Y, and W-135 antibody persistence and booster response were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group
Number analyzed (Participants) | 41 | 63 | 61
Percentage of participants
  Serogroup A; Day 0, ≥1:4 (n=41, 63, 61) | 70.7 | 76.2 | 50.8
  Serogroup A; Day 0, ≥1:8 (n=41, 63, 61) | 48.8 | 46.0 | 18.0
  Serogroup A; Day 30, ≥1:4 (n=40, 62, 59) | 100.0 | 100.0 | 93.2
  Serogroup A; Day 30, ≥1:8 (n=40, 62, 59) | 100.0 | 100.0 | 84.8
  Serogroup C; Day 0, ≥1:4 (n=41, 63, 61) | 29.3 | 20.6 | 9.8
  Serogroup C; Day 0, ≥1:8 (n=41, 63, 61) | 22.0 | 12.7 | 4.9
  Serogroup C; Day 30, ≥1:4 (n=41, 63, 59) | 100.0 | 98.4 | 59.3
  Serogroup C; Day 30, ≥1:8 (n=41, 63, 59) | 100.0 | 98.4 | 54.2
  Serogroup Y; Day 0, ≥1:4 (n=41, 63, 61) | 31.7 | 33.3 | 6.6
  Serogroup Y; Day 0, ≥1:8 (n=41, 63, 61) | 14.6 | 14.3 | 3.3
  Serogroup Y; Day 30, ≥1:4 (n=40, 63, 60) | 100.0 | 100.0 | 81.7
  Serogroup Y; Day 30, ≥1:8 (n=40, 63, 60) | 100.0 | 98.4 | 75.0
  Serogroup W-135; Day 0, ≥1:4 (n=41, 63, 61) | 43.9 | 49.2 | 14.8
  Serogroup W-135; Day 0, ≥1:8 (n=41, 63, 61) | 29.3 | 22.2 | 8.2
  Serogroup W-135; Day 30, ≥1:4 (n=40, 63, 60) | 100.0 | 100.0 | 83.3
  Serogroup W-135; Day 30, ≥1:8 (n=40, 63, 60) | 100.0 | 98.4 | 73.3

2. Other Pre Specified Outcome: Geometric Mean Antibody Titers to Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®.
Description: Antibody titers to meningococcal serogroups A, C, Y, and W-135 were measured by serum bactericidal assay using human complement (SBA-HC).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Meningococcal Serogroups A, C, Y, and W-135 Geometric Mean Titers were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group
Number analyzed (Participants) | 41 | 63 | 61
Titers (1/dilutions)
  Serogroup A; Day 0 (N=41, 63, 61) | 6.2 [4.4 to 8.8] | 7.4 [5.4 to 10.2] | 3.5 [2.9 to 4.3]
  Serogroup A; Day 30 (N=40, 62, 59) | 200.9 [134.2 to 300.6] | 234.1 [162.4 to 337.4] | 15.6 [11.7 to 20.9]
  Serogroup C; Day 0 (N=41, 63, 61) | 4.4 [2.6 to 7.3] | 2.9 [2.3 to 3.6] | 2.2 [2.0 to 2.4]
  Serogroup C; Day 30 (N=41, 63, 59) | 606.3 [422.1 to 870.9] | 397.5 [283.9 to 556.6] | 9.5 [6.2 to 14.6]
  Serogroup Y; Day 0 (N=41, 63, 61) | 3.0 [2.3 to 3.7] | 3.1 [2.5 to 3.9] | 2.1 [2.0 to 2.3]
  Serogroup Y; Day 30 (N=40, 63, 60) | 530.1 [374.4 to 750.4] | 264.6 [193.6 to 361.7] | 13.5 [9.6 to 18.9]
  Serogroup W-135; Day 0 (n=41, 63, 61) | 4.1 [3.0 to 5.8] | 3.7 [3.0 to 4.5] | 2.5 [2.1 to 2.9]
  Serogroup W-135; Day 30 (N=40, 63, 60) | 332.0 [200.1 to 550.8] | 256.0 [180.8 to 362.5] | 14.9 [10.5 to 21.3]

3. Other Pre Specified Outcome: Percentage of Participants Experiencing Solicited Injection-Site or Systemic Reactions Following Vaccination With Menactra®
Description: Solicited injection-site: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Vomiting, Drowsiness, Anorexia, Irritability, Arthralgia, and Diarrhea. Grade 3 Solicited Injection-site: Pain - Incapacitating, unable to perform usual activities; Erythema and Swelling - ≥2.0 in. Grade 3 Solicited systemic: Fever (Temperature) ->39.0˚C (>102.2˚F); Headache - Prevents daily activities; Vomiting - ≥3 episodes per 24 hours; Drowsiness - Disabling, dozing off or falling asleep while engaged in usual activities; Anorexia - Skips ≥3 meals; Irritability - >3 hours duration; Arthralgia - Unwilling to move due to pain; and Diarrhea - ≥ 5 episodes per 24 hours.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group
Number analyzed (Participants) | 48 | 66 | 67
Percentage of participants
  Injection-site Pain (N=47, 66, 65) | 55.3 | 65.2 | 63.1
  Grade 3 Injection-site Pain (N=47, 66, 65) | 2.1 | 1.5 | 0.0
  Injection-site Erythema (N=47, 66, 65) | 23.4 | 39.4 | 38.5
  Grade 3 Injection-site Erythema (N=47, 66, 65) | 6.4 | 6.1 | 15.4
  Injection-site Swelling (N=47, 66, 65) | 19.1 | 30.3 | 32.3
  Grade 3 Injection-site Swelling (N=47, 66, 65) | 8.5 | 3.0 | 12.3
  Fever (N=47, 66, 65) | 12.8 | 6.1 | 4.6
  Grade 3 Fever (N=47, 66, 65) | 0.0 | 0.0 | 0.0
  Headache (N=47, 66, 65) | 8.5 | 10.6 | 6.2
  Grade 3 Headache (N=47, 66, 65) | 2.1 | 0.0 | 0.0
  Vomiting (N=47, 66, 65) | 6.4 | 1.5 | 3.1
  Grade 3 Vomiting (n=47, 66, 65) | 0.0 | 1.5 | 1.5
  Drowsiness (N=47, 66, 65) | 19.1 | 24.2 | 10.8
  Grade 3 Drowsiness (N=47, 66, 65) | 0.0 | 0.0 | 0.0
  Anorexia (n=47, 66, 65) | 4.3 | 12.1 | 18.5
  Grade 3 Anorexia (N=47, 66, 65) | 0.0 | 0.0 | 1.5
  Irritability (N=47, 66, 65) | 19.1 | 30.3 | 33.8
  Grade 3 Irritability (N=47, 66, 65) | 2.1 | 1.5 | 4.6
  Arthralgia (n=47, 66, 65) | 8.5 | 13.6 | 16.9
  Grade 3 Arthralgia (N=47, 66, 65) | 2.1 | 1.5 | 0.0
  Diarrhea (N=47, 66, 65) | 8.5 | 10.6 | 9.2
  Grade 3 Diarrhea (N=47, 66, 65) | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 30 post-vaccination.
Arm/Group | One-Dose Menactra Group | Two-Dose Menactra Group | Menactra-naïve Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/66 | 0/67
Other Adverse Events (participants affected / at risk) | 26/48 | 43/66 | 41/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | One-Dose Menactra Group (N=48) | Two-Dose Menactra Group (N=66) | Menactra-naïve Group (N=67)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 1 (1)
Injection-site Pain (General disorders) | 26/47 (26) | 43 (43) | 41/65 (41)
Injection-site Erythema (General disorders) | 11/47 (11) | 26 (26) | 25/65 (25)
Injection-site Swelling (General disorders) | 9/47 (9) | 20 (20) | 21/65 (21)
Fever (General disorders) | 6/47 (6) | 4 (4) | 3/65 (3)
Headache (Nervous system disorders) | 4/47 (4) | 7 (7) | 4/65 (4)
Vomiting (Gastrointestinal disorders) | 3/47 (3) | 1 (1) | 2/65 (2)
Drowsiness (Nervous system disorders) | 9/47 (9) | 16 (16) | 7/65 (7)
Anorexia (Metabolism and nutrition disorders) | 2/47 (2) | 8 (8) | 12/65 (12)
Irritability (Psychiatric disorders) | 9/47 (9) | 20 (20) | 22/65 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4/47 (4) | 9 (9) | 11/65 (11)
Diarrhea (Gastrointestinal disorders) | 4/47 (4) | 7 (7) | 6/65 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications